CLINICAL TRIAL: NCT01077102
Title: Eccentric Training as Novel Rehabilitation for COPD
Brief Title: Eccentric Exercise Training as Novel Rehabilitation for Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jean Bourbeau, Jean Bourbeau, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUHC Pilot Project 2007
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema
Keywords: COPD; eccentric exercise training; cycle ergometer; muscle function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eccentric exercise training (Experimental)
  Interventions: Other: Eccentric exercise training
- Concentric exercise training (Active Comparator)
  Interventions: Other: Eccentric exercise training

INTERVENTIONS:
Other: Eccentric exercise training — The eccentric exercise training will be performed using a specially built cycle ergo meter where the pedals are driven in backward direction by an electric motor, which has to overcome the adjustable resistance of the electromagnetic brake. During eccentric cycle ergometry patients have to resist the turning pedals.

SUMMARY:
The main purpose of this project is to establish the additional value of eccentric versus concentric exercise to optimize muscle function in patients with severe COPD. With this pilot project the investigators expect that an eccentric endurance training protocol adapted to severe COPD patients will lead to gains in muscle strength, the primary outcome, and cellular adaptation (muscle morphology and oxidative capacity, mitochondrial respiratory capacity) when compared to a concentric training approach.

This information will be essential if the investigators want to design and power a randomized clinical trial that will allow assessing effectiveness of this novel rehabilitation approach.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major respiratory illness that is both preventable and treatable. Dyspnea is the most important symptom that COPD patients experience and this can have a major impact on their daily live. While COPD is characterized by a spectrum of disease severity, most patients experience poor exercise intolerance attributable to ventilatory limitation as well as peripheral muscle fatigue, ultimately leading to severe disability.

Endurance exercise is an important component of pulmonary rehabilitation and is aimed at preventing this decline in functional capacity. The effects of pulmonary rehabilitation are largely attributable to the exercise training component involving concentric muscle contractions, traditionally trough dynamic, large muscle exercise on a cycle ergometer or treadmill. However, many patients are unable to partake and benefit from such rehabilitation because of locomotor muscle weakness and severe ventilatory limitation that prevent them from exercising at intensities sufficient to provoke improvements in cardioventilatory and skeletal muscle function. Eccentric exercise is known for its unique physiologically fundamental characteristics: the lower metabolic demand for a same power output and greater muscle gains compared to the concentric exercise. For this reason, eccentric endurance training has been proposed as a novel adjunctive rehabilitative countermeasure for certain chronic diseases (such as coronary disease and COPD) and can play an important role for patients with advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* male patients with severe COPD (FEV1/FVC < 0.70 and FEV1 ≤ 50% predicted of normal)
* Patients aged 40 to 80 years old in whom exercise is not contraindicated
* Current and ex-smokers
* Patients who do not require oxygen therapy

Exclusion Criteria:

* Patients presenting neurological or orthopedic problems, morbid obesity, acute medical condition or recent exacerbations (in the last four weeks)
* Patients with recent or current participation in a rehabilitation program

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Muscle strength | At baseline, at the middle way point of the training program (5th to 7th week) and at the end of the 10-wk training program
  This outcome will be measured using an isokinetic dynamometer

SECONDARY OUTCOMES:
Muscle cellular adaptation | At baseline and at the end of the training program
  Muscle biopsy will include evaluation of cross-sectional area, fiber type, mitochondrial oxidative capacity, mitochondrial respiratory capacity, respiratory oxygen species and expression of genes involved in muscle atrophy and hypertrophy (Atrogin-1, MurF1, FoxO, MyoD, Myostatin)
Exercise capacity (maximal and submaximal) | At baseline, at the middle way point of the training program (5th to 7th week) and at the end of the 10-wk training program
Physical Activity | At baseline, at the middle way point of the training program (5th to 7th week) and at the end of the 10-wk training program
  Physical activity levels will be measured by an accelerometer and by the CHAMPS questionnaire.
Health-related quality of life (HRQL) | At baseline, at the middle way point of the training program (5th to 7th week) and at the end of the 10-wk training program
  The HRQL will be measured by the Chronic Respiratory Questionnaire
Muscle pain and creatine kinase(CK)levels | Muslce pain will be assessed in the beginning and in the end of each session and CK levels at baseline, after the fisrt week of training, midway through and the after the last week of training

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourbeau, M.D, M.Sc., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Tanja Taivassalo, Ph.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Helene Perrault, Ph.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada